CLINICAL TRIAL: NCT06716073
Title: Long-Term Outcomes of Endoscopic-assisted vs Conventional Breast-conserving Surgery in Breast Cancer Patients After Neoadjuvant Therapy: a Randomized, Multicenter, Open Label, Non-inferiority Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-648-01
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Invasive
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic breast-conserving surgery (E-BCS) group (Experimental)
  Interventions: Procedure: Surgery
- Conventional breast-conserving surgery (C-BCS) group (No Intervention)

INTERVENTIONS:
Procedure: Surgery — comparison of 2 surgical procedures
  Arms: Endoscopic breast-conserving surgery (E-BCS) group

SUMMARY:
With the title of "Long-Term Outcomes of endoscopic-assisted vs conventional breast-conserving surgery in breast cancer patients after neoadjuvant therapy: a randomized, multicenter, open label, non-inferiority trial", this study targets breast cancer patients after neoadjuvant therapy. A total of 1380 eligible patients, after screening with inclusion and exclusion criteria, will be randomly assigned to Endoscopic-assisted breast conserving surgery(E-BCS) or conventional breast conserving surgery (C-BCS) group at a 1:1 ratio using stratified block randomization method, stratified by centers and molecular subtype. The co-primary endpoints are 5-year disease-free survival (5y-DFS) and Breast-Q score at 6 months after surgery. The secondary endpoints are cosmetic outcomes including surgeons' satisfaction with breast and patients' satisfaction with scar, survival outcomes including 5-year overall survival (5y-OS) and 5-year local-recurrence rate (5y-LRR), surgical outcomes including operative time, intraoperative blood loss, incision length and postoperative complications rate. This study aims to confirm the long-term safety and aesthetic outcome of endoscopic-assisted surgery in breast cancer patients after neoadjuvant treatment by comparing it with conventional open breast conserving surgery, and provide clinical evidence for the popularized application of endoscopic breast surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18 to 75 years
2. Pathologically confirmed invasive breast cancer
3. Receiving preoperative chemotherapy (Each molecular subtype corresponds to unanimous regimen)
4. cT1-3N0-3M0
5. Unilateral breast tumor
6. Eastern Cooperative Oncology Group score 0-1
7. Left Ventricular Ejection Fraction (LVEF) ≥50%
8. Leukocytes ≥ 3.0×109/L, Absolute neutrophil count ≥ 1.5×109/L, Platelets ≥ 100×109/L, Hemoglobin ≥ 90g/L, Creatinine <1.5 × institutional ULN, Total bilirubin ≤ 2.0 × institutional ULN.

Exclusion Criteria:

1. Diffusely disseminated malignant calcification foci
2. Not applicable for BCS after neoadjuvant therapy
3. Pregnancy or breastfeeding
4. Additional malignancy
5. Severe cardiopulmonary, liver or kidney dysfunction or other systemic diseases (such as uncontrolled chronic heart failure, critical hypertension or diabetes with poor blood glucose control).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2033-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
5-year disease free survival | From surgery to the end of follow-up at 5 years
  The proportion of patients remaining after excluding patients with disease recurrence, metastasis or death from the time of surgery to 5-year follow-up
Patients' satisfaction with breast | From surgery to the follow-up at 6 months
  The score of Breast-Q scale "Satisfaction with breasts" table 6 months after surgery

SECONDARY OUTCOMES:
Surgeons' satisfaction with breast | From surgery to the follow-up at 6 months
  Surgeons evaluate the cosmetic outcome of breast based on the photos before surgery and after surgery. Four ranks: Excellent (9-10 points), Good (7-8 points), Fair (5-6 points) and Poor (0-4 points) are categorized on a basis of average total score from Ueda scale
Patients satisfaction with scar | From surgery to the follow-up at 6 months
  Scar-Q scale including 3 tables about the surgical scar: appearance, symptom, psychosocial impact with total score of 100 will be used for evaluating patients satisfaction with scar
5-year overall survival | From surgery to the end of follow-up at 5 years
  The proportion of patients remaining after excluding patients who died from any cause at 5-year follow-up
5-year local-regional recurrence rate | From surgery to the end of follow-up at 5 years
  The proportion of patients with a lump found on breast, axilla, chest wall, skin or scars of surgery ipsilateral to the surgical side through physical examination or imaging, confirmed as the same pathological type as the primary tumor according to biopsy at 5-year follow up
Postoperative complication rate | From surgery to the follow-up at 12 months
  The proportion of patients with postoperative complications including hemorrhage, incision dehiscence, upper limb lymphedema, infection,seroma.
Surgical duration | Intraoperative
  The time from the beginning of surgery to the end of surgery
Intraoperative blood loss | Intraoperative
  The blood loss during the operation
Incision length | Intraoperative
  The length of surgical incision

CONTACTS AND LOCATIONS:
Overall Officials: Shicheng Su, Doctor, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University Shenzhen Shantou Central Hospital, Shantou, Guangdong

IPD SHARING:
Plan to Share IPD: No